CLINICAL TRIAL: NCT05140356
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Neural Mechanisms and Cognitive Functions of Children With Autism Spectrum Disorder
Brief Title: Therapeutic Intervention Effects of rTMS on Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Huafu Chen, professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-chenhuafulab-003
Record Dates: First submitted 2021-11-03; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Autism
Keywords: autism; Brain Plasticity; transcranial magnetic stimulation; Magnetic Resonance Imaging; eye movement; gut microbiome
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High amplitude repeated transcranial magnetic stimulation (Experimental): Applied high amplitude repeated transcranial magnetic stimulation
  Interventions: Device: Applied high amplitude repeated transcranial magnetic stimulation
- Low amplitude repeated transcranial magnetic stimulation (Experimental): Applied low amplitude repeated transcranial magnetic stimulation
  Interventions: Device: Applied low amplitude repeated transcranial magnetic stimulation
- healthy control group (No Intervention): No intervention

INTERVENTIONS:
Device: Applied high amplitude repeated transcranial magnetic stimulation — Each mode required 20 stimuli(100%RMT) for 20 minutes each time, 5 times a week
  Arms: High amplitude repeated transcranial magnetic stimulation
Device: Applied low amplitude repeated transcranial magnetic stimulation — Each mode required 20 stimuli(15%RMT) for 20 minutes each time, 5 times a week
  Arms: Low amplitude repeated transcranial magnetic stimulation

SUMMARY:
Autism spectrum disorder (ASD) is a common and complex neurodevelopmental disorder, which is characterized by impairments of social communication, social reciprocity, as well as restricted and repetitive behaviors (RRB). The unclear pathogenesis of ASD, its increasing prevalence, and its poor clinical diagnosis and treatment effect have caused a serious economic and mental burden on patients and their families. As a new non-invasive neuroelectrophysiological technique, transcranial magnetic stimulation (TMS) has been used more and more in the interventional treatment of autism. The current project aims to explore the influence of TMS on brain plasticity in autism by using TMS for interventional treatment of autism and provide guidelines for the intervention and treatment of autism by evaluating the efficiency of these methods.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a common and complex neurodevelopmental disorder, which is characterized by impairments of social communication, social reciprocity, as well as restricted and repetitive behaviors (RRB). The unclear pathogenesis of ASD, its increasing prevalence, and its poor clinical diagnosis and treatment effect have caused a serious economic and mental burden on patients and their families. As a new non-invasive neuroelectrophysiological technique, transcranial magnetic stimulation (TMS) has been used more and more in the interventional treatment of autism. The current project aims to explore the influence of TMS on brain plasticity in autism by using TMS for interventional treatment of autism and provide guidelines for the intervention and treatment of autism by evaluating the efficiency of these methods. Investigators conduct a randomized, double-blind, controlled TMS trial and collect the participants' stool samples and sequence the gut microbiome before the first magnetic resonance imaging(MRI) scan. Besides, investigators collect brain imaging data, eye movement data and clinical scale score before and after TMS trial to explore the changes of TMS treatment on clinical behavior and brain plasticity and provide guidelines for the intervention and treatment of autism.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 2 to 8 years old. Clinical DSM-IV diagnosis of autism.

Exclusion Criteria:

* Subjects with other neurodevelopmental diseases Subjects with contraindications to MRI.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The gray matter volume of children with autism at baseline and after repeated transcranial magnetic stimulation intervention as assessed by magnetic resonance imaging. | through study completion, an average of 1 year
  Longitudinal study of the gray matter volume will be conducted in children with autism at baseline and after repeated transcranial magnetic stimulation intervention based on structural magnetic resonance image. Longitudinal effect of repeated transcranial magnetic stimulation intervention on brain structure in children with autism will be assessed by Voxel-based morphometry analysis for gray matter volume changes.

SECONDARY OUTCOMES:
The functional connectivity of whole brain of whole brain in children with autism with repeated transcranial magnetic stimulation intervention as assessed by functional magnetic resonance imaging. | through study completion, an average of 1 year
  Longitudinal study of the functional connectivity will be conducted in children with autism at baseline and after repeated transcranial magnetic stimulation intervention based on resting-state functional magnetic resonance image

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided